CLINICAL TRIAL: NCT07171619
Title: A Phase 1, Single-Sequence, 3 Period Crossover, Open-Label Study to Determine the Effect of Rabeprazole or H2 Blocker Famotidine on the Pharmacokinetics of Nirogacestat in Healthy Adult Male Participants
Brief Title: Evaluate the Effects of Famotidine or Rabeprazole on the PK of Nirogacestat
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: SpringWorks Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: NIR-DT-107
Record Dates: First submitted 2025-08-07; First posted 2025-09-12 (Actual); Last update posted 2025-09-12 (Actual); Status verified 2025-09

CONDITIONS: Healthy
MeSH Terms: interventions — nirogacestat; Amyloid Precursor Protein Secretases; Famotidine; Histamine H2 Antagonists; Rabeprazole; Proton Pump Inhibitors

STUDY DESIGN:
Intervention Model Description: Three period Crossover
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Period 1 - Nirogacestat Dose (Reference) (Active Comparator): Nirogacestat will be administered, after at least a 10-hour fast, in the morning on Day 1, Day 6, and Day 17
  Interventions: Drug: Nirogacestat
- Period 2 - Nirogacestat and Famotidine (Test) (Active Comparator): Famotidine will be administered as an oral tablet 2 hours after the administration of nirogacestat on Day 6.
  Interventions: Drug: Nirogacestat and Famotidine
- Period 3 Nirogacestat and Rabeprazole (Test) (Active Comparator): Rabeprazole will be administered as an oral tablet in the evenings on Day 10 through Day 16.
  Interventions: Drug: Nirogacestat and Rabeprazole

INTERVENTIONS:
Drug: Nirogacestat — oral dose of 150 mg nirogacestat
  Other Names: PF-03084014- GS (gamma secretase) inhibitor
  Arms: Period 1 - Nirogacestat Dose (Reference)
Drug: Nirogacestat and Famotidine — oral dose of 150 mg nirogacestat & oral dose of 40 mg famotidine
  Other Names: Histamine H2-Receptor Antagonist (H2 Blocker)
  Arms: Period 2 - Nirogacestat and Famotidine (Test)
Drug: Nirogacestat and Rabeprazole — oral dose of 150 mg nirogacestat and oral dose of 20 mg rabeprazole
  Other Names: Proton Pump Inhibitor (PPI)
  Arms: Period 3 Nirogacestat and Rabeprazole (Test)

SUMMARY:
This study will evaluate the effects of the H2 blocker famotidine or the PPI rabeprazole on the PK of nirogacestat in healthy male participants

DETAILED DESCRIPTION:
This is a phase 1, single-center, single-sequence crossover study to compare the PK, safety, and tolerability of nirogacestat alone or coadministered with famotidine or rabeprazole. This study will consist of 3 periods: Period 1 Nirogacestat Alone (Reference), Period 2 Nirogacestat and Famotidine (Test), and Period 3 Nirogacestat and Rabeprazole (Test).

There will be a screening period of up to 28 days prior to Day 1. Eligible participants will be enrolled in the study and will complete a 21-day Treatment Period. A follow-up (FU) telephone call will be performed approximately 26 days after discharge from the clinical research unit (CRU) on Day 47 (+2 days).

During screening, participants will sign the informed consent form (ICF) prior to any study procedures being performed. Participants must satisfy all the inclusion and exclusion criteria to be eligible for study participation. Participants will be admitted to the CRU on Day -1 for check-in procedures and eligibility confirmation. Participants will remain domiciled at the CRU until Day 21 after the last PK sample is collected and safety evaluations are completed.

Participants will receive a single 150 mg dose of nirogacestat in the morning of Day 1 following an overnight fast of at least 10 hours once eligibility is confirmed. Study treatment (nirogacestat) will be administered by mouth (PO) followed by 240 mL of water; otherwise, additional fluids will be restricted from 1 hour predose until 2 hours postdose. A mouth check will be done to ensure the study treatment has been consumed. Participants will continue to fast for approximately 4 hours after administration of study treatment.

On Day 6, participants will be administered a single 150 mg dose of nirogacestat in the morning after an overnight fast of at least 10 hours. Study treatment (nirogacestat) will be administered PO followed by 240 mL of water; otherwise, additional fluids will be restricted from 1 hour predose until 2 hours postdose. Two hours after the administration of nirogacestat, participants will be administered 40 mg of famotidine PO followed by 240 mL of water; additional fluids will be restricted until 2 hours post dose of famotidine and participants will continue to fast for approximately 2 hours after administration of famotidine.

Beginning in the evening of Day 10 through Day 16, participants will be administered a single dose of rabeprazole each evening. On Day 17, following an overnight fast of at least 10 hours, participants will receive a single dose of nirogacestat in the morning. Study treatment will be administered PO followed by 240 mL of water; additional fluids will be restricted from 1 hour predose until 2 hours postdose; otherwise, participants will continue to fast for approximately 4 hours after administration of nirogacestat.

Participants will remain domiciled at the CRU until all safety evaluations are completed on Day 21.

Participants will complete a FU telephone visit on Day 47 (+2 days) for review of AEs/SAEs and concomitant medications.

ELIGIBILITY:
Inclusion Criteria:

1. Participant understands the study procedures, is willing to comply with all study requirements and restrictions, and agrees to participate in the study by providing written informed consent as described in Appendix 1 of the protocol, prior to any study-related procedures being performed.
2. Participant is a male (assigned at birth) between 18 and 55 years of age (inclusive) at the time of informed consent.
3. Participant has a body mass index (BMI) ≥18.0 kg/m2 and ≤32.0 kg/m2 (inclusive) at Screening and a total body weight >50 kg.
4. Participant is considered to be medically healthy, as determined by a responsible and experienced investigator, based on a clinical evaluation (including medical history, physical examination, clinical laboratory tests, vital sign measurements, and a 12-lead ECG performed, and the results of clinical chemistry, hematology, coagulation, and urinalysis carried out at Screening and Day -1.
5. Participant has alanine aminotransferase (ALT), aspartate aminotransferase (AST), and total bilirubin levels <1.5 × the upper limit of normal (ULN) at Screening and at Day -1.
6. Participant has normal renal function (creatinine clearance ≥90 mL/min) as evidenced by normal estimated glomerular filtration rate (eGFR) measured by the CKD-EPI equation.
7. Participant agrees to the following during the treatment periods and for at least 7 days after the last dose of study treatment:

   1. Refrain from donating or preserving sperm; PLUS either
   2. Be abstinent from heterosexual intercourse as their preferred and usual lifestyle (abstinent on a long-term and persistent basis) and agree to remain abstinent.

      OR
   3. Must agree to use a male condom when having sexual intercourse with women of childbearing potential (WOCBP). An additional form of contraception should also be used by the female partner if she is of childbearing potential.
8. Has sufficiently good venous access in at least one arm to confidently enable serial blood sampling.

Exclusion Criteria:

1. Participant has a history or presence of oncologic, cardiovascular, pulmonary, hepatic, renal, hematologic, gastrointestinal, ocular, endocrine, immunologic, dermatologic, musculoskeletal, neurologic, psychiatric, or other disease or condition or laboratory test abnormality that in the investigator's judgment poses a significant risk to the safety of the participant or the achievement of study objectives.
2. Participant has a history or presence of any condition possibly affecting drug absorption (e.g., gastrectomy).
3. Participant has a medical history or abnormal findings at Screening or Day -1 that the investigator judges may put at risk achieving the objectives of the study or protecting the safety of the participant.
4. Participant has an acute illness with symptom or treatment that has started or persisted within 14 days prior to study treatment administration unless mild in severity and enrollment is approved by both investigator and sponsor's medical monitor.
5. Participant has tested positive for active Helicobacter pylori (H. pylori) infection.
6. Participant has tested positive for hepatitis B virus (HBV), hepatitis C virus (HCV), or human immunodeficiency virus (HIV) or has a clinically significant infection.
7. Participant has blood pressure (BP) that is ≥140 mmHg systolic or 90 mmHg diastolic following at least 5 minutes of rest in the supine position at Screening and Day -1. Additionally, BP that is <90 mmHg systolic or 45 mmHg diastolic following at least 5 minutes of rest at Screening and Day -1.
8. Participant has heart rate (HR) that is <40 bpm or >100 bpm after resting in a supine position for 5 minutes at Screening and Day -1.
9. Participant has averaged QT interval corrected using Fridericia formula (QTcF) results from valid triplicate ECGs >450 msec at Screening and Day -1.
10. Participant has family history of long QT syndrome or of unexplained sudden death or drowning in a first-degree relative under age 50.
11. Participant has an ECG waveform abnormality that interferes with QT/QTc interval measurement or interpretation. A participant with mild sinus arrhythmia or sparse isolated premature ventricular contractions (PVC) is eligible at the investigator's discretion.
12. Participant has a positive alcohol breath test, positive cotinine test, or other positive drug screen test at Screening or Day -1.
13. Participant has a positive nasopharyngeal rapid antigen test for SARS-CoV-2 on Day -1 or has had any known close contact with a person who tested positive for SARS-CoV-2 or with a COVID-19 patient within 2 weeks prior to admission.
14. Participant has received any vaccine within 14 days prior to the first dose of study treatment administration on Day 1.
15. Participant has received any CYP3A4 inhibitors or inducers within 21 days or 5 half-lives (whichever is longer) prior to Day 1.
16. Participant has had concurrent use of long-acting gastric acid-reducing agents within 21 days of Day 1, including H2 blockers and PPIs, including over-the-counter agents.
17. Participant has received any prescription or non-prescription drugs (including vitamins and dietary or herbal supplements), within 3 weeks or 5 half-lives, if known (whichever is longer) prior to study treatment administration on Day 1.
18. Participant has received an investigational product within 30 days or 5 times the half-lives, if known, of any drug used in the prior study (whichever is longer), or exposure to more than 3 new investigational agents within 12 months prior to study treatment administration on Day 1.
19. Participant has a known hypersensitivity or intolerance to any of the study treatments, or excipients thereof, or a history of drug or other allergy that, in the opinion of the investigator or sponsor medical monitor, contraindicates their participation.
20. Participant has a history of excessive intake of alcohol, defined as an average daily intake of >3 units, or an average weekly intake of >14 units (1 unit is equivalent to 1 can or bottle [250 mL] of beer, or 1 measure [35 mL] of spirits, or 1 glass [100 mL] of wine) in the last 6 months prior to Screening.
21. Participant has a history of illicit drug abuse within the past 2 years prior to Screening.
22. Participant has consumed red wine or any fruit juices (including but not limited to Seville oranges, grapefruit, grapefruit juice, star fruit, star fruit juice, pomelos, exotic citrus fruits, grapefruit hybrids) within 72 hours of Day -1, as outlined in Section 5.3.1.
23. Participant has used caffeine or other xanthine-containing products (e.g., coffee, black tea, green tea, colas, cacao, guarana, guayusa, yerba mate) within 24 hours of Screening and Day -1.
24. Participant regularly consumes excessive amounts (defined as >5 cups per day) of caffeine, xanthine-containing products, or energy drinks as judged by the investigator.
25. Participant has used tobacco- or nicotine-containing products within 2 months prior to Screening.
26. Participant has donated blood or had a loss of >450 mL of blood within 60 days or donation of plasma within 7 days prior to Screening.
27. Participant has received blood products within the 60 days prior to Screening.
28. Participant is unwilling to avoid strenuous or unaccustomed activity, sunbathing, or contact sports within 48 hours prior to admission to the CRU and until discharge from the CRU.
29. Participant is deemed unsuitable for this study in the opinion of the investigator for any additional reason, condition, or prior therapy.

Ages: 18 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Estimated)
Dates: Start 2025-09-09 (Actual); Primary Completion 2025-11 (Estimated); Study Completion 2025-11 (Estimated)

PRIMARY OUTCOMES:
Area under the concentration-time curve from time zero to infinity of nirogacestat. | Serial blood samples will be collected to determine concentrations of nirogacestat (in serum) on Day 1, Day 6, and Day 17 predose (-30 minutes) and 0.5, 1, 1.5, 2, 3, 4, 6, 8, 10, 12, 24, 36, 48, 72, and 96 hours postdose
  Serum AUCinf of nirogacestat.
Maximum serum concentration (Cmax) of nirogacestat. | Serial blood samples will be collected to determine concentrations of nirogacestat (in serum) on Day 1, Day 6, and Day 17 predose (-30 minutes) and 0.5, 1, 1.5, 2, 3, 4, 6, 8, 10, 12, 24, 36, 48, 72, and 96 hours postdose
  Serum Cmax of nirogacestat.
Effect of a single 2-hour staggered dose of famotidine on the PK AUCinf of nirogacestat | Serial blood samples will be collected to determine concentrations of nirogacestat (in serum) on Day 1, Day 6, and Day 17 predose (-30 minutes) and 0.5, 1, 1.5, 2, 3, 4, 6, 8, 10, 12, 24, 36, 48, 72, and 96 hours postdose
  Serum AUCinf of nirogacestat.
Effect of a single 2-hour staggered dose of famotidine on the PK Cmax of nirogacestat | Serial blood samples will be collected to determine concentrations of nirogacestat (in serum) on Day 1, Day 6, and Day 17 predose (-30 minutes) and 0.5, 1, 1.5, 2, 3, 4, 6, 8, 10, 12, 24, 36, 48, 72, and 96 hours postdose
  Serum Cmax of nirogacestat.

SECONDARY OUTCOMES:
Determine the effect of rabeprazole or famotidine on nirogacestat PK (AUClast) Area under the concentration-time curve from zero to the time last quantifiable concentration | Serial blood samples will be collected to determine concentrations of nirogacestat (in serum) on Day 1, Day 6, and Day 17 predose (-30 minutes) and 0.5, 1, 1.5, 2, 3, 4, 6, 8, 10, 12, 24, 36, 48, 72, and 96 hours postdose
  Serum AUClast
Determine the effect of rabeprazole or famotidine on nirogacestat PK (Tmax) time of maximum concentration | Serial blood samples will be collected to determine concentrations of nirogacestat (in serum) on Day 1, Day 6, and Day 17 predose (-30 minutes) and 0.5, 1, 1.5, 2, 3, 4, 6, 8, 10, 12, 24, 36, 48, 72, and 96 hours postdose
  Serum Tmax
Determine the effect of rabeprazole or famotidine on nirogacestat PK (T1/2) Terminal elimination half-life | Serial blood samples will be collected to determine concentrations of nirogacestat (in serum) on Day 1, Day 6, and Day 17 predose (-30 minutes) and 0.5, 1, 1.5, 2, 3, 4, 6, 8, 10, 12, 24, 36, 48, 72, and 96 hours postdose
  Serum T1/2
Determine the effect of rabeprazole or famotidine on nirogacestat PK (CL/F) apparent clearance after oral dose | Serial blood samples will be collected to determine concentrations of nirogacestat (in serum) on Day 1, Day 6, and Day 17 predose (-30 minutes) and 0.5, 1, 1.5, 2, 3, 4, 6, 8, 10, 12, 24, 36, 48, 72, and 96 hours postdose
  Serum CL/F
Determine the effect of rabeprazole or famotidine on nirogacestat PK (Vd/F) Apparent oral volume of distribution | Serial blood samples will be collected to determine concentrations of nirogacestat (in serum) on Day 1, Day 6, and Day 17 predose (-30 minutes) and 0.5, 1, 1.5, 2, 3, 4, 6, 8, 10, 12, 24, 36, 48, 72, and 96 hours postdose
  Serum Vd/F
To evaluate the Adverse Events in healthy male participants after a single 150 mg dose of nirogacestat administered with and without rabeprazole or famotidine | Baseline through Day 21 and includes the Follow-up Phone Call
  Safety assessments will include assessments of all adverse events (AEs) including any serious adverse events (SAEs) and graded using the most current version of the Common Terminology Criteria for Adverse Events CTCAE Version 5.0 condition-specific scale
Number of Participants with Clinical Laboratory Tests Values Outside the Normal Reference Range | Baseline (Day -1) through Day 21.
  The laboratory test includes assessment of chemistry, hematology, coagulation, and urinalysis based on Investigator's decision/assessment.
To evaluate the vital sign measurements in healthy male participants after a single 150 mg dose of nirogacestat administered with and without rabeprazole or famotidine | Baseline (Day -1) through Day 21.
  Safety assessments will include assessments of all vital sign measurements of Heart Rate, Blood Pressure, Respirations and Body Temperature
To evaluate ECG parameters in healthy male participants after a single 150 mg dose of nirogacestat administered with and without rabeprazole or famotidine | Baseline (Day -1) through Day 21.
  Safety assessments will include assessments of all electrocardiograms (ECGs) to include heart rate and measures PR, QRS, QT, and QTcF and QT corrected using Bazett's formula (QTcB).
To evaluate physical examination findings in healthy male participants after a single 150 mg dose of nirogacestat administered with and without rabeprazole or famotidine | Baseline (Day -1) through Day 21.
  Safety assessments will include assessments of all physical examination findings to include assessments of the cardiovascular, dermatological, respiratory, gastrointestinal, skin, and neurological systems

CONTACTS AND LOCATIONS:
Overall Officials: Mary Beth Brune, MD, Principal Investigator — Medpace, Inc.
Locations (1):
- Medpace, Cincinnati, Ohio, United States

IPD SHARING:
Plan to Share IPD: Yes
SpringWorks Therapeutics is committed to data transparency and sharing data to further research while maintaining the privacy and confidentiality of research participants. Pertinent participant-level data from completed clinical trials will be made available by SpringWorks to qualified researchers upon approval of reasonable requests following de-identification/anonymization pursuant to applicable law.